CLINICAL TRIAL: NCT04451330
Title: A Multi-Center, Randomized, Double-Blind, Placebo Controlled Study To Compare Efficacy and Safety of Trifarotene (CD5789) Cream When Used Withan Oral Antibiotic for the Treatment of Severe Acne Vulgaris
Brief Title: A Study to Compare Efficacy and Safety of Trifarotene Cream When Used With an Oral Antibiotic for the Treatment of Severe Acne Vulgaris (AV)
Acronym: DUAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.202394
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2021-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — trifarotene; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trifarotene Cream + Doxycycline (Experimental): Participants were applied with Trifarotene (CD5789) 50 micrograms per gram (mcg/g) cream topically on the face once daily in the evening for 12 weeks and received doxycycline 120 milligrams (mg) tablet orally once daily in the evening and 1 tablet in the morning on Day 2 of every week for 12 weeks.
  Interventions: Drug: Trifarotene cream; Drug: Doxycycline hyclate
- Trifarotene Vehicle + Doxycycline Placebo (Placebo Comparator): Participants were applied with vehicle CD5789 topically on the face once daily in the evening for 12 weeks and received doxycycline matching placebo tablet orally once daily in the evening and 1 tablet in the morning on Day 2 of every week for 12 weeks.
  Interventions: Drug: Trifarotene Vehicle; Drug: Doxycycline Placebo

INTERVENTIONS:
Drug: Trifarotene cream — Trifarotene 50 mcg/g cream applied topically once daily on face for 12 weeks.
  Other Names: AKLIEF
  Arms: Trifarotene Cream + Doxycycline
Drug: Doxycycline hyclate — Doxycycline hyclate delayed release 120 mg tablets was administered orally for 12 weeks.
  Other Names: DORYX MPC
  Arms: Trifarotene Cream + Doxycycline
Drug: Trifarotene Vehicle — Trifarotene 50 mcg/g vehicle cream was applied topically once daily on face for 12 weeks.
  Arms: Trifarotene Vehicle + Doxycycline Placebo
Drug: Doxycycline Placebo — Doxycycline hyclate delayed release 120 mg placebo tablets was administered orally for 12 weeks.
  Arms: Trifarotene Vehicle + Doxycycline Placebo

SUMMARY:
The purpose of this study was to demonstrate that daily use of topical trifarotene (CD5789) 50 microgram per gram (mcg/g) cream when used in association with oral antibiotic is safe and effective for the treatment of severe AV.

ELIGIBILITY:
Inclusion Criteria:

* Participants with clinical diagnosis of acne vulgaris, defined by IGA score of 4 (Severe)
* Participants with at least 20 inflammatory lesions (papules and pustules) and 30 to 120 non-inflammatory lesions (open comedones and closed comedones) and no more than 2 nodules (less than [<]1 centimeter [cm] in diameter) on the face, excluding the nose
* Agrees to provide written informed consent
* Participant is a female of non-childbearing potential (premenarchal or postmenopausal [absence of menstrual bleeding for 1 year prior to Screening, without any other medical reason], hysterectomy or bilateral oophorectomy)

Exclusion Criteria:

* Participant with any acne cyst on the face
* Participants with nodulocystic or conglobate acne, acne fulminans, or secondary acne (chloracne, drug-induced acne, etc.)
* Participants with facial dermal conditions (example [e.g.] tattoo, skin abrasion, eczema, sunburned skin, scars, nevi, etc.) that may interfere with study assessments in the opinion of the investigator
* Participants who is at risk in terms of precautions, warnings, and contraindications for trifarotene or doxycycline hyclate
* Currently receiving any prescription testosterone therapy (e.g., testosterone cypionate, testosterone enanthate, testosterone pellet, testosterone undecanoate) or on a testosterone booster or prescription testosterone (e.g., dehydroepiandrosterone [DHEA], Omnadren, Sustanon, testosterone cypionate, testosterone enanthate, testosterone propionate, testosterone phenylpropionate) or testosterone supplements (e.g., Tribulus).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (24):
  - Galderma Investigational Site, Fort Smith, Arkansas
  - Galderma Investigational Site, Hot Springs, Arkansas
  - Galderma Investigational Site, Rogers, Arkansas
  - Galderma Investigational Site, Newport Beach, California
  - Galderma Investigational Site, Aventura, Florida
  - Galderma Investigational Site, Boca Raton, Florida
  - Galderma Investigational Site, Miramar, Florida
  - Galderma Investigational Site, Newnan, Georgia
  - Galderma Investigational Site, Evansville, Indiana
  - Galderma Investigational Site, New Albany, Indiana
  - Galderma Investigational Site, Rockville, Maryland
  - Galderma Investigational Site, Warren, Michigan
  - Galderma Investigational Site, New Brighton, Minnesota
  - Galderma Investigational Site, Las Vegas, Nevada
  - Galderma Investigational Site, Stony Brook, New York
  - Galderma Investigational Site, High Point, North Carolina
  - Galderma Investigational Site, Sugarloaf, Pennsylvania
  - Galderma Investigational Site, Charleston, South Carolina
  - Galderma Investigational Site, Knoxville, Tennessee
  - Galderma Investigational Site, Arlington, Texas
  - Galderma Investigational Site, Dallas, Texas
  - Galderma Investigational Site, Grapevine, Texas
  - Galderma Investigational Site, Pflugerville, Texas
  - Galderma Investigational Site, San Antonio, Texas
- Galderma Investigational Site, Aibonito, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at United States of America and Puerto Rico between 29 Jul 2020 and 26 Apr 2021.
Pre-assignment Details: A total of 202 participants were randomized in 2:1 ratio in 2 treatment groups.
Groups:
- Trifarotene (CD5789) Cream + Doxycycline: Participants were applied with Trifarotene (CD5789) 50 micrograms per gram (mcg/g) cream topically on the face once daily in the evening for 12 weeks and received doxycycline 120 milligrams (mg) tablet orally once daily in the evening and 1 tablet in the morning on Day 2 of every week for 12 weeks.
Period: Overall Study
Arm/Group | Trifarotene (CD5789) Cream + Doxycycline | Trifarotene Vehicle + Doxycycline Placebo
Started | 133 | 69
Completed | 123 | 65
Not Completed | 10 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 5 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Withdrawal by parent/guardian | 1 | 0
Not completed — Other than specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent to treat (ITT) population that included all participants who were randomized.
Groups:
- Trifarotene + Doxycycline: Participants were applied with Trifarotene (CD5789) 50 micrograms per gram (mcg/g) cream topically on the face once daily in the evening for 12 weeks and received doxycycline 120 milligrams (mg) tablet orally once daily in the evening and 1 tablet in the morning on Day 2 of every week for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Trifarotene + Doxycycline | Trifarotene Vehicle + Doxycycline Placebo | Total
Number analyzed (Participants) | 133 | 69 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.0 (7.30) | 20.3 (8.92) | 20.1 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 43 | 123
  Male | 53 | 26 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 20 | 70
  Not Hispanic or Latino | 83 | 49 | 132
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 6 | 15
  White | 114 | 58 | 172
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Facial Total Lesions Counts [Mean (Standard Deviation); unit: Lesion counts] — Total lesion counts corresponded to the sum of inflammatory and non-inflammatory lesions, and papules. The investigator (or subinvestigator) counted all inflammatory lesions (papules, pustules, and nodular lesions) and noninflammatory lesions (open and closed comedos; diagnosis based on palpation) on the face.
  Lesion counts | 101.5 (40.11) | 100.7 (33.91) | 101.2 (38.02)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Facial Total Lesion Counts to Week 12
Description: Total lesion counts corresponded to the sum of inflammatory and non-inflammatory lesions, and papules. The investigator (or subinvestigator) counted all inflammatory lesions (papules, pustules, and nodular lesions) and non-inflammatory lesions (open and closed comedos; diagnosis based on palpation) on the face.
Time Frame: From Baseline to Week 12
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (Standard Deviation); unit: Lesion counts
Arm/Group | Trifarotene + Doxycycline | Trifarotene Vehicle + Doxycycline Placebo
Number analyzed (Participants) | 133 | 69
Lesion counts | -69.1 (2.28) | -48.1 (3.14)

2. Secondary Outcome: Absolute Change From Baseline in Facial Inflammatory Lesions (IL) Counts to Week 12
Description: All inflammatory lesions (papules, pustules, and nodular lesions) were counted by investigator/subinvestigator.
Time Frame: From Baseline to Week 12
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: Lesion counts
Arm/Group | Trifarotene + Doxycycline | Trifarotene Vehicle + Doxycycline Placebo
Number analyzed (Participants) | 133 | 69
Lesion counts | -29.4 (1.09) | -19.5 (1.49)

3. Secondary Outcome: Absolute Change From Baseline in Facial Non Inflammatory Lesions (NIL) Counts to Week 12
Description: Non-inflammatory lesions (open and closed comedo) were counted by investigator/subinvestigator.
Time Frame: From Baseline to Week 12
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (Standard Deviation); unit: Lesion counts
Arm/Group | Trifarotene + Doxycycline | Trifarotene Vehicle + Doxycycline Placebo
Number analyzed (Participants) | 133 | 69
Lesion counts | -39.5 (1.42) | -28.2 (1.96)

4. Secondary Outcome: Percentage of Participants Who Achieved an IGA Score of 1 (Almost Clear) or 0 (Clear) and At Least a 2-Grade Improvement From Baseline to Week 12
Description: IGA was an assessment scale used to evaluate facial acne severity. IGA was recorded from components collected on the case report form (CRF) using a 5-point scale where (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on inflammation, pustules and papulation/infiltration. Success Rate was defined as the percentage of participants who achieved an IGA score of 1 (Almost Clear) or 0 (Clear) and at least a 2-grade improvement from Baseline to Week 12.
Time Frame: From Baseline to Week 12
Population: The ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Trifarotene + Doxycycline | Trifarotene Vehicle + Doxycycline Placebo
Number analyzed (Participants) | 133 | 69
percentage of participants | 31.7 | 15.8

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 12.
Description: Analysis was performed on safety population which comprised of all randomized participants who applied/took the study drug at least once.
Arm/Group | Trifarotene + Doxycycline | Trifarotene Vehicle + Doxycycline Placebo
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/133 | 0/69
Other Adverse Events (participants affected / at risk) | 0/133 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trifarotene + Doxycycline (N=133) | Trifarotene Vehicle + Doxycycline Placebo (N=69)
Self-Injurious Ideation (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04451330/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT04451330/SAP_001.pdf